CLINICAL TRIAL: NCT02472054
Title: First Line Treatment of Familiar Lymphohistiocytosis by Alemtuzumab (CAMPATH®)
Brief Title: Treatment of Familiar Lymphohistiocytosis
Acronym: C-HLH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P120109; 2014-005585-30 (EudraCT Number)
Record Dates: First submitted 2015-06-08; First posted 2015-06-15 (Estimated); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Hemophagocytic Lymphohistiocytosis (HLH)
Keywords: hemophagocytic lymphohistiocytosis (HLH); Alemtuzumab (CAMPATH®)
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — Alemtuzumab; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- hemophagocytic lymphohistiocytosis (HLH) (Experimental): Alemtuzumab (CAMPATH®)
  1. Initial Treatment (D1 to D3) D1: 0.5 mg / kg / day Alemtuzumab combined with 2 mg /kg/d of IV Methylprednisolone (MP) or PO Prednisolone, and IVC or PO cyclosporine (CSA) (target rate from 150 to 200 ng / ml in the absence of renal failure) D2 and D3: 1 mg / kg / day Alemtuzumab combined with 2 mg / kg / d of IV MP or PO Prednisolone and IVC or PO CSA (target rate 150-200 ng / ml)
     The maximum dose of Alemtuzumab is limited to 30 mg per day (1 vial).
  2. Maintenance treatment (D4 to D14)
     * MP/Prednisolone progressive tapering starting at D4 (2 mg / kg / day) to reach the dose 0.5 mg / kg / day at D14
     * CSA IVC or PO at a target rate of 150-200 ng / ml
  Interventions: Drug: Alemtuzumab; Drug: Methyl Prednisolone (MP); Drug: Cyclosporin A (CSA)

INTERVENTIONS:
Drug: Alemtuzumab
  Other Names: CAMPATH®
Drug: Methyl Prednisolone (MP)
Drug: Cyclosporin A (CSA)

SUMMARY:
The purpose of this project is to study the number of surviving patients until hematopoietic stem cell transplantation (HSCT) after first line treatment of hemophagocytic lymphohistiocytosis (HLH) by Alemtuzumab

DETAILED DESCRIPTION:
The hemophagocytic lymphohistiocytosis (HLH) or lymphohistiocytic activation syndrome is an inflammatory condition caused by a uncontrolled proliferation of activated lymphocytes and macrophages secreting an excess of inflammatory cytokines. Familial hemophagocytic lymphohistiocytosis (FHL) is a rare disorder of the immune system, which is invariably fatal when untreated. Treatment requires the achievement of remission of HLH prior to allogeneic hematopoietic stem cell transplantation, the only curative therapy to date.

Despite significant progress in the treatment, mortality remains high and an important number of patients will die before being eligible for HSCT.

A better understanding of the pathophysiology of FHL has opened new avenues for immunotherapy. Based on previous observations concerning the utilization of Anti-thymoglobulins (ATG) for the treatment of patients with FHL, the protocol propose a new therapeutic strategy using Alemtuzumab in association with steroids as first line treatment in FHL. This proposition is based on the hypothesis that Alemtuzumab, capable of killing T lymphocytes efficiently in vivo, should be better tolerated than ATG. In fact, in contrast to the mechanism of action of ATG, Alemtuzumab does not activate T lymphocytes.

A better tolerance and efficacy of Alemtuzumab is expected in the treatment of the hemophagocytic lymphohistiocytic syndrome. This may have a positive impact not only on survival until HSCT, but also on overall survival and quality of life with regard to long-term neurological sequelae.

This is a multicenter, open, phase I/II, non-comparative, non randomized study. Patients are recruited by the investigators during hospitalization for a first episode of lymphohistiocytic activation syndrome requiring specific treatment.

Several visits (including the final visit) are scheduled within the trial over a period of approximately 10 months for all patients, from the signature of the consent up to 6 months after hematopoietic stem cell transplantation.

The recruitment period will be 48 months; the total period of the study is 58 months. The treatment consists in an intravenous administration of CAMPATH®.

For the research purpose, investigators will collect specific samples for:

* biobank (Cytokine dosage) at the inclusion visit and the day prior to the conditioning;
* pharmacokinetics of CAMPATH® : at every cure of CAMPATH® and every week. Also diagnostic lumbar puncture at the inclusion visit, day 14 is required to document the response to treatment and to determine the result of the therapeutic care.

The efficacy of the treatment will be measured to Day14, Day21 and Day28. All adverse events must be reported in the e-Case Report Form (e-CRF)

ELIGIBILITY:
Inclusion Criteria :

* Patient < 18 years
* Patient with diagnosis of hemophagocytic lymphohistiocytic syndrome confirmed by at least one of the following two criteria :

  * Genetic diagnosis FHL or other genetic disease predisposing to HLH like Chediak-Higashi syndrome, Griscelli syndrome type II and X-linked lymphoproliferative syndrome type I and II (XLP-1 and XLP-2) or positive family history of HLH
  * Presence of at least 5 of the following 8 criteria (diagnostic criteria as defined by the "Histiocyte Society" ) :
  * Fever
  * Splenomegaly
  * Cytopenia (affecting at least two cell lineages : Hemoglobin <9.0 g / dl, Platelets <100.000/μl, Absolute neutrophil count (ANC) <1.000/µl)
  * Hypertriglyceridemia and / or hypofibrinogenemia (Fasting triglycerides ≥ 3 mmol / l, Fibrinogen ≤ 1.5 g / l)
  * Haemophagocytosis found in a histological specimen (without evidence of a malignant process and rheumatic disease)
  * Decreased or absent NK function (<10% of the laboratory standard)
  * Ferritin ≥ 500μg / l
  * Soluble CD25 ≥ 2.400U/ml or presence of activated T cells in the immune phenotyping
* Patient without prior specific treatment of lymphohistiocytic activation syndrome or under treatment with corticosteroids and / or ciclosporin.
* Patient beneficiary of a health insurance scheme
* Holder (s) of parental authority who signed the informed consent
* Man or woman in reproductive age willing to take reliable contraceptive measures during the treatment and 6 months after the end of the treatment

Specific situation of patients with neurological involvement :

Most patients with neurological involvement caused by a HLH will meet the inclusion criteria. However some patients may present an isolated neurological involvement as the first manifestation of familiar lymphohistiocytosis as described in the literature. These patients do not always present all the inclusion criteria. However their clinical condition may justify their inclusion prior to the confirmation of a genetic diagnosis and/or the detection of all required diagnostic inclusion criteria.

In the absence of the required 5 out of 8 diagnostic criteria, the eventual inclusion of patients with predominant neurological involvement will be evaluated by a scientific committee to judge their inclusion or not in the study. The remaining inclusion and exclusion criteria must be fulfilled. A written report will be established.

Exclusion Criteria :

* Age ≥ 18 years
* Patients previously treated with Anti-Thymoglobulin (SAL), etoposide (VP16) or Alemtuzumab.
* Confirmed or suspected diagnosis of a malignant or rheumatic disease
* Contraindication (s) to the administration of Alemtuzumab :

  * Hypersensitivity to murine proteins or to any of the excipients (sodium chloride, dibasic sodium phosphate, potassium chloride, potassium dihydrogen phosphate, polysorbate 80, disodium edetate dihydrate, and water for injection)
  * General evolving infection except infections that are the triggering factor of the HLH .
  * HIV
  * Progressing malignant tumors
  * Pregnancy

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Number of surviving patients until HSCT | Day 1 until transplantation, up to 4 months

SECONDARY OUTCOMES:
Number of complete remissions following treatment | Day 14, Day 21, Day 28
  To assess the efficacy of the Alemtuzumab
Time of delay between the first administration of Alemtuzumab and complete remission | Day 14, Day 21, Day 28
  To assess the efficacy of the Alemtuzumab
Dosage of Alemtuzumab | Day1-3, Day7, Day15-16, Day22-23, Day28
  Pharmacokinetic
Number of side effects | Day 1 until transplantation, up to 4 months
  To assess the tolerance of the Alemtuzumab

CONTACTS AND LOCATIONS:
Overall Officials: Alain FISCHER, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No